CLINICAL TRIAL: NCT01084083
Title: A Phase II Trial of Induction Chemotherapy Followed by Cetuximab (Erbitux) With Low Dose vs. Standard Dose IMRT in Patients With HPV-Associated Resectable Squamous Cell Carcinoma of the Oropharynx
Brief Title: Induction Chemotherapy Followed By Cetuximab and Radiation in HPV-Associated Resectable Stage III/IV Oropharynx Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000665170; ECOG-E1308 (Other: Eastern Cooperative Oncology Group); U10CA023318 (NIH)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer; Precancerous Condition
Keywords: human papilloma virus infection; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Precancerous Conditions; Papillomavirus Infections; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Cetuximab; Radiotherapy, Intensity-Modulated; Paclitaxel; Albumin-Bound Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): After induction therapy with Paclitaxel and Cisplatin, patients undergo low-dose intensity-modulated radiotherapy (IMRT) 5 days per week for approximately 5 weeks (27 fractions). Patients also receive cetuximab IV over 1-2 hours once weekly for 6 weeks.
  Interventions: Biological: cetuximab; Radiation: intensity-modulated radiation therapy (IMRT); Drug: Paclitaxel; Drug: Cisplatin
- Group 2 (Experimental): After induction therapy with Paclitaxel and Cisplatin, patients undergo standard-dose IMRT 5 days per week for approximately 6 weeks (33 fractions). Patients also receive cetuximab IV over 1-2 hours once weekly for 7 weeks.
  Interventions: Biological: cetuximab; Radiation: intensity-modulated radiation therapy (IMRT); Drug: Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Biological: cetuximab — Given IV
Radiation: intensity-modulated radiation therapy (IMRT) — Patients undergo low-dose OR standard dose IMRT based on their clinical response to induction therapy
Drug: Paclitaxel — Given IV, 90 mg/m^2 on days 1, 8 and 15
  Other Names: Abraxane, Taxol
Drug: Cisplatin — Given IV, 75 mg/m^2 on day 1
  Other Names: Platinol

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high energy x-rays to kill tumor cells. Giving paclitaxel, cisplatin, and cetuximab together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying paclitaxel, cisplatin, and cetuximab to see how well they work when followed by cetuximab and two different doses of intensity-modulated radiation therapy in treating patients with HPV-associated stage III or stage IV cancer of the oropharynx that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of induction therapy comprising paclitaxel, cisplatin, and cetuximab followed by cetuximab in combination with low-dose or standard-dose intensity-modulated radiotherapy, as measured by 2-year progression-free survival (PFS), in patients with human papillomavirus(HPV)-associated resectable stage III-IVB squamous cell carcinoma of the oropharynx.

Secondary

* To assess overall survival.
* To evaluate the objective response, local control, and metastatic rate.
* To evaluate early and late toxicities of treatment.

Tertiary

* To evaluate quality of life and speech and swallowing function as measured by Functional Assessment of Cancer Therapy - General (FACT-G), Functional Assessment of Cancer Therapy-Head and Neck (FACT-HN), and Vanderbilt Head and Neck Symptom Survey (VHNSS).
* To assess the effect of treatment-induced fatigue on general physical functioning in patients with head and neck cancer.
* To correlate functional decline with clinical, physical, and biologic correlatives.
* To evaluate radiation-resistance markers, including ERCC1 single nucleotide polymorphism and protein expression, and to correlate them with treatment efficacy.
* To demonstrate the usefulness of biomarkers, including ERCC1, epidermal growth factor receptor (EGFR), cytokine and chemokine markers, and plasma transforming growth factor alpha (TGFA) and transforming growth factor beta (TGFB) levels, in predicting progression-free survival (PFS) and other outcome parameters.
* To evaluate the correlation between the efficacy of cetuximab and polymorphisms in FcγR-receptors.
* To evaluate functional outcome and biological parameters, including telomere length, angiotensin-converting enzyme polymorphism, and C-reactive protein level.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive cisplatin intravenously (IV) over 1 hour on day 1 and paclitaxel IV over 3 hours and cetuximab IV over 1-2 hours on days 1, 8, and 15. Treatment repeats every 21 days for 3 courses. Patients then undergo evaluation of response to induction therapy. Patients with a clinical complete response (CR) at the primary tumor site proceed to group 1 of concurrent radiotherapy and cetuximab. Patients with a clinical partial response (PR) or stable disease (SD) at the primary tumor site or those with grossly positive disease at the primary tumor site proceed to group 2 of concurrent radiotherapy and cetuximab.
* Concurrent radiotherapy and cetuximab: Treatment begins 14-21 days after the last day of induction therapy.

  * Group 1 (CR): Patients undergo low-dose intensity-modulated radiotherapy (IMRT) 5 days per week for approximately 5 weeks (27 fractions). Patients also receive cetuximab IV over 1-2 hours once weekly for 6 weeks.
  * Group 2 (PR, SD, or grossly positive disease): Patients undergo standard-dose IMRT 5 days per week for approximately 6 weeks (33 fractions). Patients also receive cetuximab IV over 1-2 hours once weekly for 7 weeks.

Patients complete questionnaires assessing fatigue, physical function, weight loss, quality of life, head and neck symptom burden, and speech and swallowing function at baseline and at 1, 6, 12, and 24 months after completion of study treatment.

Tumor tissue and serum samples may be collected periodically for correlative laboratory studies.

After completion of study treatment, patients are followed up periodically for 3 years.

PROJECTED ACCRUAL: 83 patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the oropharynx as determined by Hematoxylin and eosin (H&E) staining

  * Newly diagnosed disease
  * Resectable disease OR disease that is expected to become resectable after study treatment
  * Stage III, IVA, or IVB disease as determined by imaging studies (computed tomography (CT) scan with IV contrast or magnetic resonance imaging (MRI) required) and a complete head and neck exam
* Paraffin-embedded tumor specimen available for central confirmation of HPV-associated disease as determined by H&E staining and in-situ hybridization (ISH) for HPV-16 and immunohistochemistry (IHC) for p16

  * HPV-associated disease is defined as p16 IHC-positive and/or HPV-16 ISH-positive
  * Non-HPV-associated disease is defined as p16 IHC-negative
  * NOTE: If there is limited tumor material, p16 IHC will be performed before HPV-16 ISH
* Measurable disease of the primary tumor or nodes by clinical and radiographic methods, defined as a lesion that is ≥ 2 cm in at least one dimension by clinical exam AND by radiographic exam with CT scan or MRI (or a lesion that is ≥ 1 cm in at least one dimension if the radiographic exam utilizes spiral CT scan)
* No primary tumor or nodal metastasis fixed to the carotid artery, skull base, or cervical spine
* No evidence of distant metastases
* Eastern Cooperative Oncology Group performance status 0-1
* Granulocytes ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Total serum bilirubin ≤ 1.5 mg/dL
* Creatinine clearance ≥ 60 mL/min
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of another malignancy (except for carcinoma in situ of the cervix and/or nonmelanomatous skin cancer) unless it has been curatively treated and the patient has been disease-free for ≥ 2 years
* Patients with any of the following within the past 6 months are eligible provided they have been evaluated by a cardiologist and/or neurologist before study entry:

  * New York Heart Association (NYHA) class III-IV congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Unstable angina
  * Myocardial infarction (with or without ST elevation)

Exclusion Criteria:

* Prior chemotherapy
* Prior radiotherapy above the clavicles
* Prior surgery with curative intent for this disease (complete head and neck exam with biopsy allowed)
* Prior therapy specifically and directly targeting the EGFR pathway
* Prior severe infusion reaction to a monoclonal antibody
* Uncontrolled diabetes, uncontrolled infection despite antibiotics, or uncontrolled hypertension within the past 30 days
* Concurrent illness likely to interfere with study therapy or to prevent surgical resection
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-08-11 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanthi Marur, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (121):
- United States (121):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - California Cancer Care, Incorporated - Greenbrae, Greenbrae, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford Cancer Center, Stanford, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Evanston Hospital, Evanston, Illinois
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Stony Brook University Cancer Center, Stony Brook, New York
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Franklin, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin

REFERENCES:
- [Result] Marur S, Li S, Cmelak AJ, Gillison ML, Zhao WJ, Ferris RL, Westra WH, Gilbert J, Bauman JE, Wagner LI, Trevarthen DR, Balkrishna J, Murphy BA, Agrawal N, Colevas AD, Chung CH, Burtness B. E1308: Phase II Trial of Induction Chemotherapy Followed by Reduced-Dose Radiation and Weekly Cetuximab in Patients With HPV-Associated Resectable Squamous Cell Carcinoma of the Oropharynx- ECOG-ACRIN Cancer Research Group. J Clin Oncol. 2017 Feb 10;35(5):490-497. doi: 10.1200/JCO.2016.68.3300. Epub 2016 Dec 28. PMID 28029303
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on March 17, 2010, accrued its first patient on August 11, 2010, and closed to accrual on October 19, 2011, with an accrual of 90 patients from 16 ECOG-affiliated institutions.
Groups:
- Overall: Patients receive cisplatin IV on day 1 and paclitaxel IV and cetuximab IV on days 1, 8, and 15. Treatment repeats every 21 days for 3 courses. Patients then undergo evaluation of response to induction therapy. Patients with a CR at the primary tumor site proceed to group 1 of concurrent low-dose IMRT and cetuximab. Patients with a PR or SD at the primary tumor site or those with grossly positive disease at the primary tumor site proceed to group 2 of concurrent standard dose IMRT and cetuximab.
Period: Overall Study
Arm/Group | Overall
Started | 90
Treated | 89 (This is the all treated patients for toxicity analysis)
Eligible | 81
Eligible and Treated | 80 (This is the eligible and treated patients for secondary efficacy endpoints)
CR to Induction Therapy | 56
CR and Treated With 5400 cGy IMRT | 44 (This is the primary study population for the primary endpoint (24-month PFS).)
Completed | 78
Not Completed | 12
Not completed — Adverse Event | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Complicating disease | 1
Not completed — Other | 2
Not completed — Never started assigned therapy | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Eligible and Treated Patients: Patients receive cisplatin IV on day 1 and paclitaxel IV and cetuximab IV on days 1, 8, and 15. Treatment repeats every 21 days for 3 courses. Patients then undergo evaluation of response to induction therapy. Patients with a CR at the primary tumor site proceed to group 1 of concurrent low-dose IMRT and cetuximab. Patients with a PR or SD at the primary tumor site or those with grossly positive disease at the primary tumor site proceed to group 2 of concurrent standard dose IMRT and cetuximab.
Arm/Group | Eligible and Treated Patients
Number analyzed (Participants) | 80
Age, Continuous [Median (Full Range); unit: Years] | 57 [35 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 76
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: 24-month Progression-free Survival
Description: 24-month progression-free survival is defined as the proportion of patients who were alive and progression-free at 24 months post registration. The primary study population for this endpoint is patients who were confirmed post-induction clinical complete response (CR) at their primary sites and subsequently received 5400 cGy radiation therapy to their primary sites.
Time Frame: assessed within 14 days after delivery of the third cycle of induction therapy, and 8 weeks and 6 months after completion of concurrent therapy, then every 6 months until progression or until 3 years from study entry
Population: patients who were confirmed post-induction clinical complete response (CR) at their primary sites and subsequently received 5400 cGy radiation therapy to their primary sites
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Primary Study Population: The primary study population for this endpoint is patients who were confirmed post-induction clinical complete response (CR) at their primary sites and subsequently received 5400 cGy radiation therapy to their primary sites.
Arm/Group | Primary Study Population
Number analyzed (Participants) | 44
percentage of participants | 64 [48 to 78]

2. Secondary Outcome: 24-months Overall Survival
Description: OS was defined as the time from registration to death, or censored at last date known alive. Kaplan-Meier method was used to estimate the overall survival rate at 24 months.
Time Frame: as for outcome 1
Population: eligible and treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eligible and Treated Patients
Number analyzed (Participants) | 80
percentage of participants | 91 [82 to 96]

3. Secondary Outcome: Primary Clinical Response Rate
Description: Primary clinical response rate is defined as the proportion of patients with complete response or partial response at their primary sites after induction therapy. Response status for the primary site was classified by clinical examination using endoscopy. If, however, the clinical response status of the primary was unclear based on endoscopy, then the CT or MRI (required at the end of induction) was used to determine status of the primary. If clinical and radiological evaluation of the primary was unclear, a biopsy was considered at the discretion of the treating physician.
Time Frame: assessed within 14 days after delivery of the third cycle of induction therapy
Population: eligible and treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eligible and Treated Patients
Number analyzed (Participants) | 80
percentage of participants | 73 [61 to 82]

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment and for 3 months after completion of concurrent treatment to capture late radiation toxicities
Groups:
- All Treated Patients: Patients receive cisplatin IV on day 1 and paclitaxel IV and cetuximab IV on days 1, 8, and 15. Treatment repeats every 21 days for 3 courses. Patients then undergo evaluation of response to induction therapy. Patients with a CR at the primary tumor site proceed to group 1 of concurrent low-dose IMRT and cetuximab. Patients with a PR or SD at the primary tumor site or those with grossly positive disease at the primary tumor site proceed to group 2 of concurrent standard dose IMRT and cetuximab.
  Adverse events data were reported for all patients received at least one dose of protocol therapy.
Arm/Group | All Treated Patients
Serious Adverse Events (participants affected / at risk) | 69/89
Other Adverse Events (participants affected / at risk) | 86/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Patients (N=89)
Tinnitus (Ear and labyrinth disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Fatigue (General disorders) | 7
Pain (General disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 29
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 20
Mucositis oral (Gastrointestinal disorders) | 29
Nausea (Gastrointestinal disorders) | 8
Oral pain (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Anorectal infection (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 9
Wound complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Cardiac troponin I increased (Investigations) | 1
CD4 lymphocytes decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 18
Neutrophil count decreased (Investigations) | 10
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Renal and urinary disorders - Other (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Patients (N=89)
Anemia (Blood and lymphatic system disorders) | 14
Fatigue (General disorders) | 45
Alopecia (Skin and subcutaneous tissue disorders) | 39
Dry skin (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash acneiform (Skin and subcutaneous tissue disorders) | 64
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 36
Dysphagia (Gastrointestinal disorders) | 27
Mucositis oral (Gastrointestinal disorders) | 50
Nausea (Gastrointestinal disorders) | 32
Oral pain (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 8
Dermatitis radiation (Injury, poisoning and procedural complications) | 23
Lymphocyte count decreased (Investigations) | 14
Neutrophil count decreased (Investigations) | 15
Weight loss (Investigations) | 31
White blood cell decreased (Investigations) | 23
Anorexia (Metabolism and nutrition disorders) | 29
Dehydration (Metabolism and nutrition disorders) | 12
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 16
Dysgeusia (Nervous system disorders) | 26
Peripheral sensory neuropathy (Nervous system disorders) | 13
Sore throat (Respiratory, thoracic and mediastinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less